CLINICAL TRIAL: NCT03863821
Title: Effects of Heated Humidified High-Flow Nasal Cannula During Six-Minute Walk Test in Patient With COPD Undergoing Pulmonary Rehabilitation
Brief Title: The Application and Analysis of HHHFNC in Walking Test of Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PL-201808008-M
Record Dates: First submitted 2019-03-04; First posted 2019-03-05 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-11

CONDITIONS: COPD; Pulmonary Disease; Rehabilitation
Keywords: chronic obstructive pulmonary disease; heated humidified high-flow nasal cannula; pulmonary rehabilitation; six-minute walking test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Intervention Model Description: Participants with COPD who done pulmonary function test will enroll to this study. Left-side heart failure, COPD AE within 3 months, diagnosed neuromuscular disease, and unable to perform 6-MWT will be exclude.
  Participants will received HHHNFC or non-HHHFNC support during the 6-MWT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HHHFNC group (Experimental): Practice 6 MWT with HHHFNC
  Interventions: Device: HHHFNC
- non-HHHFNC group (No Intervention): Practice 6 MWT without HHHFNC

INTERVENTIONS:
Device: HHHFNC — HHHFNC setting:
  1. Flow rate: 40L/min
  2. FiO2: 0.4
  HHHFNC will use immediately before 6MWT and remove at the end of 6MWT
  Arms: HHHFNC group

SUMMARY:
The aim of this study is to investigate the use heated humidified high-flow nasal cannula (HHHFNC) in pulmonary rehabilitation and analysis of cardiopulmonary parameters in adult patients.

DETAILED DESCRIPTION:
Objectives： The aim of this study is to investigate the use heated humidified high-flow nasal cannula (HHHFNC) in pulmonary rehabilitation and analysis of cardiopulmonary parameters in adult patients.

Background： Recently, HHHFNC has been used in both adult and neonates with post-extubation respiratory support. Studies indicate that HHHFNC has similar efficacy compared to non-invasive positive pressure ventilation and superior than conventional oxygen therapy. Six-minute walking test (6-MWT) is a standardized laboratory tests to evaluate the endurance capacity in adult patients. It helps clinician to modify the treatment plan. Cirio, et at. has been shown HHHFNC may improve the exercise performance in severe chronic obstructive pulmonary disease (COPD) patients with ventilatory limitation.

Study Design： This is a prospective clinical trial in a pulmonary rehabilitation out-patient department (2018.08.01-2019.07.31).。 Methods： Patents with COPD who done pulmonary function test will enroll to this study. Left-side heart failure, COPD acute-exacerbation (AE) within 3 months, diagnosed neuromuscular disease, and unable to perform 6-MWT will be exclude. The data will be collected for and analyzed.

Effect： Investigators expect the exercise performance; cardiopulmonary function will be improve under HHHFNC support. We hope the application of HHHFNC in adult patient with pulmonary rehabilitation could enhance the quality of life.

Key words： chronic obstructive pulmonary disease; heated humidified high-flow nasal cannula; pulmonary rehabilitation, six-minute walking test.

ELIGIBILITY:
Inclusion Criteria:

* COPD with performed pulmonary function test

Exclusion Criteria:

* Left-side heart failure
* COPD exacerbation within 3 month
* Diagnosed neuromuscular disease
* Unable to perform 6-MWT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-18 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Walking distance | 6 minutes
  Meter

SECONDARY OUTCOMES:
Heart rate | 1 hour
  beat per minute
Oxygen saturation (SpO2) | 1 hour
Transcutaneous carbon dioxide (PtcCO2) | 1 hour
  mmHg
Cardiac output by non-invasive cardiometry | 1 hour
  mL
Borg dyspnea scale | 1 hour
  0-10 level (level 10 means worst)

CONTACTS AND LOCATIONS:
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cirio S, Piran M, Vitacca M, Piaggi G, Ceriana P, Prazzoli M, Paneroni M, Carlucci A. Effects of heated and humidified high flow gases during high-intensity constant-load exercise on severe COPD patients with ventilatory limitation. Respir Med. 2016 Sep;118:128-132. doi: 10.1016/j.rmed.2016.08.004. Epub 2016 Aug 8. PMID 27578482
- [Result] Maltais F, Singh S, Donald AC, Crater G, Church A, Goh AH, Riley JH. Effects of a combination of umeclidinium/vilanterol on exercise endurance in patients with chronic obstructive pulmonary disease: two randomized, double-blind clinical trials. Ther Adv Respir Dis. 2014 Dec;8(6):169-81. doi: 10.1177/1753465814559209. PMID 25452426
- [Result] Man WD, Mustfa N, Nikoletou D, Kaul S, Hart N, Rafferty GF, Donaldson N, Polkey MI, Moxham J. Effect of salmeterol on respiratory muscle activity during exercise in poorly reversible COPD. Thorax. 2004 Jun;59(6):471-6. doi: 10.1136/thx.2003.019620. PMID 15170026
- [Derived] Chao KY, Liu WL, Nassef Y, Tseng CW, Wang JS. Effects of high-flow nasal cannula with oxygen on self-paced exercise performance in COPD: A randomized cross-over trial. Medicine (Baltimore). 2021 Dec 23;100(51):e28032. doi: 10.1097/MD.0000000000028032. PMID 34941043